CLINICAL TRIAL: NCT05512468
Title: Application of Preoperative Axillary Lymph Node Marking With Nano-Carbon in Breast Cancer Patients Before Neoadjuvant Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-TATOO-2020
Record Dates: First submitted 2022-08-22; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer; Neoadjuvant Therapy; Sentinel Lymph Node Biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Tattooing of biopsied node (Other): Prior to NST, suspicious axillary lymph nodes were biopsied by core needle or fne needle aspiration. The largest and/or biopsy-confrmed metastastic node was then injected with highly purifed carbon suspension either at the time of biopsy or at a separate session.
  Interventions: Drug: carbon dye

INTERVENTIONS:
Drug: carbon dye — Tattooing (marking) of biopsied node with carbon dye at the time or at a separate session of fine needle aspiration or core biopsy or separate visit under ultrasound guidance. The dye will be injected in the cortex of the node and the perinodal tissue under ultrasound guidance. Patients will undergo standard (routine) armpit surgery and may receive neoadjuvant chemotherapy as planned by the clinical team. This could be removal of a few lymph glands (sentinel node biopsy) or removal of all the lymph glands (axillary lymph node dissection) in the armpit. The surgeon will try to identify and remove the tattooed lymph gland at the time of planned armpit surgery.

SUMMARY:
The primary aim of this prospective, multicentre study is to determine whether the involved node can be marked using black carbon dye and successfully identified at the time of surgery. The secondary aims are to determine the concordance between the tattooed node and sentinel node, migration of black dye into other nodes, and false-negative rate of tattooed node (in patients undergoing ALND after NACT).

DETAILED DESCRIPTION:
Pretreatment evaluation of axillary lymph nodes and marking of biopsied nodes in patients with newly diagnosed breast cancer is becoming routine practice. Tagging of biopsied axillary lymph nodes with metal markers, similar to what is done for suspicious breast lesions, is being adopted in clinical practice. The need to mark a positive axillary lymph node becomes especially relevant in cases where neoadjuvant chemotherapy (NACT) is anticipated so that these nodes may be identified at the time of surgery. Measures that improve both the accuracy of nodal evaluation after NACT and the ability to assess treatment response are desirable in order to tailor therapies for breast cancer treatment. The investigators sought to test tattooing of biopsied axillary lymph nodes with a sterile black carbon suspension.

ELIGIBILITY:
Inclusion Criteria:

1. Female; 2. Aged >=18 years; 3. With invasive breast cancer; 4. Patients to be treated with neoadjuvant chemotherapy; 5. Patients scheduled to undergo routine fine needle aspiration (FNA) or core biopsy of abnormal axillary lymph node; 6. Patients with operable breast cancer; 7. Heart, lung, liver and kidney function well, suitable for patients undergoing surgery; 8. Informed consent patients.

Exclusion Criteria:

* 1. Patients who do not plan or are unable to operate; 2. Patients with distant metastasis were excluded; 3. Patients without invasive cancer components in DCIS alone; 4. Patients who are unable to cooperate with the doctor's recommended surgical treatment (breast conserving surgery or radical surgery) due to personal or family factors; 5. Patients with serious cardiopulmonary diseases, uncontrolled infectious diseases and other non tumor related diseases who can not tolerate comprehensive treatment such as surgery and chemotherapy; 6. Patients with mental illness or other reasons unable to sign informed consent; 7. Patients with poor medical compliance who cannot complete the trial treatment process and follow-up according to the standard according to the researcher's opinion.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Identification rate of tattooed node | 12 months
  Proportion of patients in whom tattooed node/s were identified.

SECONDARY OUTCOMES:
Concordance of tattooed node and sentinel node | 12 months
  Concordance rate: defined as the percent of patients in whomthe tattooed nodeis the sentinel node.
Migration of black dye into other nodes | 12 months
  The number of black nodes at the time of sentinel node biopsy or axillary lymph node dissection.

CONTACTS AND LOCATIONS:
Overall Officials: China Fujian, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Study Officials, Fuzhou, Fujian, China